CLINICAL TRIAL: NCT01343329
Title: Controlling Hyperadrenergic Activity in Neurologic Injury
Acronym: CHAIN
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unable to enroll subjects that fit study criteria.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Wendy Ziai, Associate Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00043058
Record Dates: First submitted 2011-04-26; First posted 2011-04-28 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Traumatic Brain Injury; Dysautonomia
Keywords: Traumatic Brain Injury; Dysautonomia; Brain Injury; Sympathetic hyperactivity
MeSH Terms: conditions — Brain Injuries, Traumatic; Autonomic Nervous System Diseases; Brain Injuries | interventions — esmolol; Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Subjects Receiving Esmolol (Experimental): The Esmolol arm is defined as a 48-hour intravenous infusion of esmolol (Brevibloc 20mg/ml), which will be started on enrollment.
  Interventions: Drug: Esmolol
- Subjects receiving Propranolol (Active Comparator): The comparison arm will be comprised of oral propranolol, starting with 20mg PO every 6 hours prn (as needed) to reduce heart rate into target range. If 20mg is ineffective, the dose will be doubled at each dosing interval until an adequate dose is found, not to exceed 120mg four times daily. (ex: 20mg, 40mg, 80mg, 120mg)
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Esmolol — The Esmolol arm is defined as a 48-hour intravenous infusion of esmolol (Brevibloc 20mg/ml), which will be started on enrollment. The infusion rate will begin at 50 micrograms/kg/min and be adjusted to achieve heart rates between 80 and 100 beats/min with standard dosing regimens used in our Neuro intensive care unit. The infusion will be started at a rate of 0.05 milligrams/kg/min (50 micrograms/kg/min) for 5 minutes. After the 5 minutes of initial infusion, maintenance infusion may be continued at 0.05 mg/kg/min or increased stepwise (e.g. 0.1 mg/kg/min, 0.15 mg/kg/min to a maximum of 0.2 mg/kg/min) with each step being maintained for 4 or more minutes until the target heart rate is achieved.
  Other Names: Brevibloc
  Arms: Subjects Receiving Esmolol
Drug: Propranolol — The comparison arm will be comprised of oral propranolol, starting with 20mg PO every 6 hours prn (as needed) to reduce heart rate into target range. If 20mg is ineffective, the dose will be doubled at each dosing interval until an adequate dose is found, not to exceed 120mg four times daily. (ex: 20mg, 40mg, 80mg, 120mg)
  Other Names: Inderal
  Arms: Subjects receiving Propranolol

SUMMARY:
Traumatic brain injury (TBI) is frequently associated with a hyperadrenergic state accompanied by elevated levels of plasma catecholamines. In its more severe presentation, the hyperadrenergic state presents as dysautonomia, which is characterized by paroxysmal alteration in vital signs, including tachycardia. The investigators hypothesize that intravenous (IV) esmolol is as effective at controlling heart rate in hyperadrenergic states as oral propranolol, which is the standard of care. Our primary endpoint is efficacy of IV esmolol vs a PRN regimen of intermittent B-blockade in controlling heart rate below a pre-specified level (< 100 bpm) after Traumatic Brain Injury (TBI) or hemorrhagic neurologic injury. Heart rates will be recorded continuously as well as hourly.

ELIGIBILITY:
Inclusion Criteria:

* TBI (Moderate/Severe TBI (GCS 12 or Head AIS>1) or hemorrhagic neurologic injury
* Hyperadrenergic Activity: At least one paroxysmal episode (lasting at least 15 minutes) of Heart Rate 110 beats per minute during two or more consecutive days plus at least two more of the following that may not be better explained by another disease process (ex: sepsis):

Temperature of 38.5C Respiratory Rate 20 breaths per minute Agitation Diaphoresis Dystonia Stimulus responsive ("triggering of paroxysm")

- Informed Consent obtained

Exclusion Criteria:

* Patients that do not meet criteria for dysautonomia (as stated above)
* Age <18 years
* Pregnancy
* Hypotension - requiring pressor therapy to maintain baseline adequate CPP or mean arterial pressure
* Cardiac arrhythmia - sinus bradycardia (HR <60), 2nd or 3rd degree AV block
* Hemodynamic contraindications to intravenous beta-blockade such as a documented history of congestive heart failure (CHF), dependency on cardiac inotropes or documented bronchospastic disease
* Any patient on chronic beta blockade as an outpatient.
* Life expectancy < 48 hours or patients with "do not resuscitate orders"
* Ongoing seizure activity
* Informed consent not obtained

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2014-02-14 (Actual); Study Completion 2014-02-14 (Actual)

PRIMARY OUTCOMES:
Controlling heart rate in traumatic brain injured patients | 72 hrs
  Once the patient is randomized and start getting the study medication, we monitor heart rate and other vital signs for 72hrs

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Ziai, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hortnagl H, Hammerle AF, Hackl JM, Brucke T, Rumpl E, Hortnagl H. The activity of the sympathetic nervous system following severe head injury. Intensive Care Med. 1980 May;6(3):169--7. doi: 10.1007/BF01757299. PMID 7391345
- [Background] Baguley IJ. Autonomic complications following central nervous system injury. Semin Neurol. 2008 Nov;28(5):716-25. doi: 10.1055/s-0028-1105971. Epub 2008 Dec 29. PMID 19115177
- [Background] Fernandez-Ortega JF, Prieto-Palomino MA, Munoz-Lopez A, Lebron-Gallardo M, Cabrera-Ortiz H, Quesada-Garcia G. Prognostic influence and computed tomography findings in dysautonomic crises after traumatic brain injury. J Trauma. 2006 Nov;61(5):1129-33. doi: 10.1097/01.ta.0000197634.83217.80. PMID 17099518
- [Background] Cotton BA, Snodgrass KB, Fleming SB, Carpenter RO, Kemp CD, Arbogast PG, Morris JA Jr. Beta-blocker exposure is associated with improved survival after severe traumatic brain injury. J Trauma. 2007 Jan;62(1):26-33; discussion 33-5. doi: 10.1097/TA.0b013e31802d02d0. PMID 17215730
- [Background] Baguley IJ, Heriseanu RE, Felmingham KL, Cameron ID. Dysautonomia and heart rate variability following severe traumatic brain injury. Brain Inj. 2006 Apr;20(4):437-44. doi: 10.1080/02699050600664715. PMID 16716989
- [Background] Meythaler JM, Stinson AM 3rd. Fever of central origin in traumatic brain injury controlled with propranolol. Arch Phys Med Rehabil. 1994 Jul;75(7):816-8. PMID 8024432
- [Background] Chiolero RL, Breitenstein E, Thorin D, Christin L, de Tribolet N, Freeman J, Jequier E, Schutz Y. Effects of propranolol on resting metabolic rate after severe head injury. Crit Care Med. 1989 Apr;17(4):328-34. doi: 10.1097/00003246-198904000-00006. PMID 2702842
- [Background] Pranzatelli MR, Pavlakis SG, Gould RJ, De Vivo DC. Hypothalamic-midbrain dysregulation syndrome: hypertension, hyperthermia, hyperventilation, and decerebration. J Child Neurol. 1991 Apr;6(2):115-22. doi: 10.1177/088307389100600204. PMID 2045626
- [Background] Silver JK, Lux WE. Early onset dystonia following traumatic brain injury. Arch Phys Med Rehabil. 1994 Aug;75(8):885-8. doi: 10.1016/0003-9993(94)90113-9. PMID 8053795
- [Background] Cuny E, Richer E, Castel JP. Dysautonomia syndrome in the acute recovery phase after traumatic brain injury: relief with intrathecal Baclofen therapy. Brain Inj. 2001 Oct;15(10):917-25. doi: 10.1080/02699050110065277. PMID 11595088
- [Background] Chen JM, Heran BS, Perez MI, Wright JM. Blood pressure lowering efficacy of beta-blockers as second-line therapy for primary hypertension. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD007185. doi: 10.1002/14651858.CD007185.pub2. PMID 20091622
- [Background] Harwood TN, Butterworth J, Prielipp RC, Royster RL, Hansen K, Plonk G, Dean R. The safety and effectiveness of esmolol in the perioperative period in patients undergoing abdominal aortic surgery. J Cardiothorac Vasc Anesth. 1999 Oct;13(5):555-61. doi: 10.1016/s1053-0770(99)90007-1. PMID 10527224
- See also: Main website for Johns Hopkins Hospital — http://www.hopkinsmedicine.org/